CLINICAL TRIAL: NCT02484339
Title: Phase II Open-label Study to Evaluate the Efficacy and Safety of Radium in Combination With External Beam Radiotherapy (EBRT) vs. EBRT Alone in the Treatment of Castration Resistant Prostate Carcinoma With Limited Bone Metastases
Brief Title: Treatment of Advanced Castration Resistant Prostate Carcinoma With Limited Bone Metastases (α-RT)
Acronym: α-RT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ursula Nestle, Prof.Dr. med, University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: α-RT
Record Dates: First submitted 2015-05-13; First posted 2015-06-29 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride; Congresses as Topic; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group A (Experimental): Radium-223 dichloride (Xofigo®) 55 kilobecquerel (kBq)/kgbw (6 i.v. injections every 4 weeks)
  External beam radiotherapy (EBRT)->conventional or high dose radiotherapy
  Interventions: Drug: Radium-223 dichloride; Other: Conventional or high dose radiotherapy
- Treatment Group B (Other): External beam radiotherapy (EBRT) ->conventional or high dose radiotherapy
  Interventions: Other: Conventional or high dose radiotherapy

INTERVENTIONS:
Drug: Radium-223 dichloride — Arm A: EBRT and timely sequential start with Radium-223 dichloride 55 kBq/kgbw (6 i.v. injections every 4 weeks) and best supportive care until progression or intolerable toxicity.
  Other Names: Xofigo®
  Arms: Treatment Group A
Other: Conventional or high dose radiotherapy — Arm B: External beam radiotherapy (EBRT)->->conventional or high dose radiotherapy
  Other Names: External beam radiotherapy (EBRT)

SUMMARY:
Phase II open-label study to evaluate the efficacy and safety of Radium-223 dichloride in combination with external beam radiotherapy (EBRT) vs. external beam radiotherapy alone in the treatment of advanced castration resistant prostate carcinoma with limited bone metastases.

To evaluate if time to radiological progression according to the "Recommendations of the Prostate Cancer Clinical Trials Working Group" published by Scher et al. (JCO 2008) (based on new lesions in bone scan and CT /MRI or death) of Radium-223 dichloride combined with EBRT is superior compared to EBRT alone.

DETAILED DESCRIPTION:
This is an international, multi-center, open-label, prospective, phase II study designed to assess the efficacy of radiation therapy in combination with Radium-223 dichloride in patients diagnosed with CRPC and oligo metastases bone disease. All patients enrolled in this study will have signed an informed consent form (ICF) and will adhere to all inclusion and exclusion criteria.

During the treatment period, patients will be followed on an ongoing basis for safety and quality of life (QoL). Safety assessments will include the collection of all AEs of any grade, serious adverse events (SAEs), adverse event (AEs) corresponding to symptoms arising from bone metastases, laboratory values, (WHO/ECOG) performance status (PS). Documentation of the date of disease progression will be performed at intervals and imaging methods (bone scans and CR/MRI) described in the study protocol. Quality of life will be measured by patient assessment using a validated questionnaire, the Brief Pain Inventory Short Form (BPI-SF), the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C15-PAL and the EORTC QLQ- Bone Metastases (BM) 22. Follow-up assessments for safety AEs and SAEs, and the occurrence of secondary malignancies will be conducted every 3-12 months until the patient dies or until the study is terminated by the sponsor. If the patient can no longer travel to the clinical site, he will be followed up for survival only, i.e., the long term follow-up phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent. Subjects must be able to understand and be willing to sign the written informed consent form (ICF). Age ≥ 18 and ≤ 85 years
2. Patients with progressive castration resistant prostate cancer (CRPC) with 1-5 bone metastases for whom Radium-223 dichloride constitutes first-line cytostatic treatment
3. Primary tumor (and its local recurrence, if applicable) controlled by effective local treatment
4. If diagnosed, pelvic lymph node metastases controlled by effective local treatment
5. At least 1 not previously locally treated skeletal metastasis on bone scan without non-bone distant metastases (e.g. lung, liver, and/or brain metastases) and without pathologically enlarged lymph nodes above the pelvis
6. Progressive disease is defined either by:

   * The appearance of new bone lesions. If progression is based on new lesion(s) on bone scan only without an increase in prostate specific antigen (PSA), PSA values from 3 assessments within the last 6 months must be provided; OR
   * In the absence of new bone lesions by 2 consecutive increases in serum PSA over previous reference value, which should not be more than 6 months before screening, each measured at least 1 week apart with the last PSA ≥5 ng/mL
7. Life expectancy of at least 6 months.
8. (WHO/ECOG) Performance Status (PS) 0 or 1
9. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to start of therapy:
10. Patient has or has had symptoms (e. g. pain or micro)

Exclusion Criteria:

Excluded medical conditions:

1. More than 5 not previously locally treated bone metastases as diagnosed by bone scintigraphy;
2. Visceral or lymph node metastases above the pelvis as assessed by computed tomography (CT) (or other imaging modality) ;
3. History of HIV infection or chronic hepatitis B or C
4. Active clinically serious infections (> grade 2 National Cancer Institute Common Terminology Criteria (NCI-CTC) version 4.03)
5. History of organ allograft
6. Patients undergoing renal dialysis
7. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study if not in complete remission for at least 5 years since date of diagnosis treated treated basal cell carcinoma, superficial bladder tumors [Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
8. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
9. Imminent or history of spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI)
10. Any other serious illness or medical condition
11. Fecal incontinence
12. Any condition that is unstable or could jeopardize the safety of the patient and his compliance in the study
13. Known allergy to Radium-223 dichloride (i.e. to active substance or one of the constituents)

Excluded therapies and medications, previous and concomitant:

1. Anticancer chemo- or targeted therapy for CRPC
2. Radiotherapy for prostate cancer manifestations other than study treatment if not given with curative intent to prostate fossa and/or pelvic lymph nodes
3. Major surgery within 4 weeks of study entry.
4. Systemic therapy with radionuclides for the treatment of bone metastases
5. Autologous bone marrow transplant or stem cell rescue within 4 months of study entry
6. Use of biologic response modifiers, such as Granulocyte-Colony Stimulating Factor (G-CSF), within 3 week of study entry
7. Investigational drug therapy outside of this trial during or within 4 weeks of study entry

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to radiological progression free survival (PFS) rate | randomization to radiological progression
  measured every 3 month by Bone Scan and MRI or CT until Follow up 7 (month 24) and after that in long term follow up every 6 month

SECONDARY OUTCOMES:
Time to local progression in any of the EBRT treated bone metastases of conventional radiotherapy (CRT) vs. High-dose image-based conformal radiotherapy (HIRT) treatment techniques | Time to local progression in any of the EBRT treated bone metastases
  measured every 3 month by Bone Scan, Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) until month 24 after that in long term follow up every 6 month with open end
Overall survival | randomization to death
  Follow up every 3 month until month 24 and after that in long term follow up every 6 month
Time to distant bone metastasis progression outside the RT target volumes | Screening to FU 7 (after 24 months) and than in long term follow up every 6 month
  Follow up every 3 month until month 24 and than in long term follow up every 6 month measured by increasing of PSA, CT/MRI
Time to Skeletal Related Event (SRE) | Screening to FU 7 (after 24 months) and than in long term follow up every 6 month
  measured every 3 month by Bone Scan, Magnetic Resonance Imaging (MRI) or Computed Tomography (CT) until month 24 and than in long term follow up every 6 month with open end
Pain control | Screening to FU 7 (after 24 months) and than in long term follow up every 6 month
  measured every 3 month by the Brief Pain Inventory Short Form (BPI-SF), the European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-C15-PAL and the EORTC QLQ- Bone Metastases (BM) 22 until month 24 and than in long term follow up every 6 month
Disease Control Rate (DCR); Response rates according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Screening to FU 7 (after 24 months) and than in long term follow up every 6 month
  Follow up every 3 month until month 24 measured by RECIST criteria and than in long term follow up every 6 month
PSA response, time to PSA response and time to PSA normalization | Screening to FU 7 (after 24 months) and than in long term follow up every 6 month
  Follow up every 3 month until month 24 and after that long term follow up every 6 month measured by PSA level
Bone alkaline phosphatase (ALP) response, time to bone ALP response | Screening to FU 7 (after 24 months) and than in long term follow up every 6 month
  Follow up every 3 month until month 24 and than long term follow up every 6 month measured by blood level

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Nestle, Principal Investigator — University Hospital Freiburg, Germany
Locations (6):
- Germany (6):
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Freiburg, Klinik für Strahlenheilkunde, Freiburg im Breisgau
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Nuklearmedizin, Mainz
  - Klinikum der Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No